CLINICAL TRIAL: NCT02134561
Title: Assessment of the Psychological, Cognitive and Social Resources of Applicants for Huntington's Disease and Presymptomatic Genetic Testing
Acronym: PREHUNT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A00088-37
Record Dates: First submitted 2014-04-10; First posted 2014-05-09 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2013-02

CONDITIONS: Presymptomatic Huntington Disease
MeSH Terms: interventions — Interview, Psychological; Neuropsychological Tests

ARMS (1):
- All subjects (Other): psychological interview, MRI, neurological tests, cognitive tests
  Interventions: Behavioral: psychological interview; Radiation: MRI; Other: cognitive tests; Other: neurological tests

INTERVENTIONS:
Behavioral: psychological interview
Radiation: MRI — This MRI is a specific intervention assign to the subjects of the study, that's why it is an interventionnal study
Other: cognitive tests
Other: neurological tests

SUMMARY:
The purpose of this study is to assess the psychological, cognitive and social resources of applicants for Huntington's Disease and Presymptomatic Testing.

ELIGIBILITY:
Inclusion Criteria:

* Applicants for Huntington's Disease and Presymptomatic Testing
* Aged 18 years and above
* Huntington disease family member
* Subject gave its written consent

Exclusion Criteria:

* No national health insurance affiliation
* Being under guardianship
* Meeting brain MRI exclusion criteria (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body, Renal failure, hypersensitivity of Gadolinium) or refusing MRI.
* Patient with movement disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline total score of the psychological Unified Huntington's Disease Rating Scale at 2 years | 3 months before diagnostic (baseline) ; 2 years after diagnostic,

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, Pays de la Loire Region, France